CLINICAL TRIAL: NCT05425147
Title: Correlation Between Perioperative Autonomic Function and Adverse Events Such as Post-induction Hypotension in Elderly Patients
Brief Title: Correlation Between Perioperative Autonomic Function and Post-induction Hypotension in Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCHanesthesia-elderly
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Intraoperative Hypotension
Keywords: post-induction hypotension, autonomic function, elderly patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-induction hypotension group: Post-induction hypotension is defined as systolic blood pressure (SBP) <90 mmHg, mean arterial pressure (MAP) <65 mmHg, or a decrease of more than 30% of baseline within 20 minutes after induction or before incision.
  Interventions: Other: Perioperative autonomic function assessment
- Stable blood pressure group: All enrolled elderly patients will undergo surgery under general anesthesia after preoperative monitoring. Those patients whose blood pressure is relatively stable after induction and does not meet the PIH criteria is classified as the stable blood pressure group.
  Interventions: Other: Perioperative autonomic function assessment

INTERVENTIONS:
Other: Perioperative autonomic function assessment — Patients will have BRS and HRV measurements taken for approximately 20 minutes, one day before surgery and on the day of surgery. We use LiDCO rapid to conduct non-invasive pulse and beat-to-beat blood pressure monitoring.

SUMMARY:
Elderly patients have a higher risk of post-induction hypotension (PIH). The decreased cardiovascular autonomic function at baseline in elderly patients may contribute to the development of PIH. The objective of our study is to effect of preoperative cardiovascular autonomic modulation in PIH, we will recruit elderly patients who are going to have general anesthesia surgery and measure preoperative baroreflex sensitivity (BRS) and heart rate variability (HRV). The primary outcome will be PIH. Secondary outcomes included: early intraoperative hypotension, postoperative complications, and 30-day postoperative mortality.

DETAILED DESCRIPTION:
With the deepening of the aging population, the number of elderly patients undergoing surgery is also increasing. These elderly patients have a declining physiological reserve and face challenges in anesthesia management: studies have shown that elderly patients are at high risk of intraoperative adverse events and postoperative complications. Post-induction hypotension (PIH) refers to the hypotension that occurs between anesthesia induction and skin incision. The current diagnostic criteria have not been fully unified. Patients with intraoperative PIH have a higher risk of postoperative death and damage to vital organs such as the heart and kidneys, and have a poor prognosis. Elderly patients are a high-risk group for PIH. Therefore, it is of great meaning to quantify the risk factors of PIH in elderly patients.

Cardiovascular autonomic function may play an essential role in intraoperative blood pressure regulation. The pressure sensor of the cardiovascular system sends the blood pressure signal to the central nervous system, and regulates the blood pressure to an appropriate level through a compensatory reflex (i.e., baroreflex). Baroreflex function can be quantified by observing the R-R interval response to an arterial blood pressure change and the results are expressed as baroreflex sensitivity (BRS). In addition to BRS, heart rate variability (HRV) can also be used to assess cardiovascular autonomic function. HRV is a promising quantitative marker of autonomic activity, which includes the time domain and frequency domain analysis of R-R interval rhythm.

Some studies have explored the relationship between preoperative cardiovascular autonomic function and PIH. However, these studies did not assess preoperative volume status, and they did not measure BRS, which is probably more connected with baroreflex.

We hypothesized that the decreased baroreflex sensitivity at baseline in elderly patients may contribute to the development of PIH. To explore the effect of preoperative cardiovascular autonomic modulation in PIH in elderly patients, we are going to measure preoperative BRS and HRV in those who were about to undergo general anesthesia surgery.

We are conducting a single-center, prospective cohort study. Elderly patients (over 65 years of age) who are going to have elective surgery under general anesthesia will be recruited and will have BRS and HRV measurements taken for approximately 20 minutes, one day before surgery and on the day of surgery. We use LiDCO rapid to conduct non-invasive pulse and beat-to-beat blood pressure monitoring. In addition to spontaneous BRS and HRV assessment, the patients will be instructed to perform round-lip breathing at 0.1 Hz for 1 minute to gain more information about BRS and HRV through respiratory sinus arrhythmia (RSA).

The primary outcome will be PIH. Secondary outcomes included: early intraoperative hypotension, postoperative complications, and 30-day postoperative mortality. Anesthesia induction medications and intraoperative monitoring data will be recorded. The intraoperative monitoring meets the standards of basic physiologic monitors recommended by American Society of Anesthesiologists (ASA). We will use Clavien-Dindo classification to describe postoperative complications. Patients will be followed up during hospitalization and 30 days after the surgery by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old;
* Elective non-cardiac surgery;
* ASA Class I-III;
* General anesthesia;
* Use a tracheal tube as an airway management tool;
* Patients and their families can understand the research protocol and are willing to participate in this research

Exclusion Criteria:

* Severe vascular disease;
* Secondary hypertension;
* Parkinson's disease;
* Cannot measure upper extremity blood pressure for various reasons;
* Arrhythmias such as atrial fibrillation cannot perform HRV measurement;
* Mentally abnormal and unable to cooperate

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients who will undergo general anesthesia surgery in Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Post-induction hypotension | within 20 minutes after induction or before incision
  Systolic blood pressure (SBP) <90 mmHg, mean arterial pressure (MAP) <65 mmHg, or a decrease of more than 30% of baseline

SECONDARY OUTCOMES:
Early intraoperative hypotension | within 30 minutes after incision
  Systolic blood pressure (SBP) <90 mmHg, mean arterial pressure (MAP) <65 mmHg, or a decrease of more than 30% of baseline
postoperative complications | 30 days after the surgery
  postoperative complications (Clavien-Dindo classification)
mortality | 30 days after the surgery
  death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Padley JR, Ben-Menachem E. Low pre-operative heart rate variability and complexity are associated with hypotension after anesthesia induction in major abdominal surgery. J Clin Monit Comput. 2018 Apr;32(2):245-252. doi: 10.1007/s10877-017-0012-4. Epub 2017 Mar 14. PMID 28293808
- [Background] Ziemssen T, Siepmann T. The Investigation of the Cardiovascular and Sudomotor Autonomic Nervous System-A Review. Front Neurol. 2019 Feb 12;10:53. doi: 10.3389/fneur.2019.00053. eCollection 2019. PMID 30809183
- [Background] La Rovere MT, Pinna GD, Raczak G. Baroreflex sensitivity: measurement and clinical implications. Ann Noninvasive Electrocardiol. 2008 Apr;13(2):191-207. doi: 10.1111/j.1542-474X.2008.00219.x. PMID 18426445
- [Derived] Cui Q, Che L, Zang H, Yu J, Xu L, Huang Y. Association between preoperative autonomic nervous system function and post-induction hypotension in elderly patients: a protocol for a cohort study. BMJ Open. 2023 Jan 30;13(1):e067400. doi: 10.1136/bmjopen-2022-067400. PMID 36717143